CLINICAL TRIAL: NCT05943730
Title: The Validity of a Seismocardiography Device to Estimate Peak Oxygen Uptake in Patients Awaiting Major Elective Surgery
Brief Title: Validity of Measuring Preoperative Fitness Using Seismofit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northumbria University (Other)
Collaborators: South Tees Hospitals NHS Foundation Trust (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); York Teaching Hospitals NHS Foundation Trust (Other); VentriJect ApS (Industry); Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1614
Record Dates: First submitted 2023-07-04; First posted 2023-07-13 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-06

CONDITIONS: Preoperative Care; Validity
Keywords: Seismocardiography; Preoperative Exercise; Peak oxygen uptake; VO2max; Cardiopulmonary exercise test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Seismofit Validity (Experimental): Participants will undergo a seismocardiography assessment, whilst supine, using the seismofit device. This will estimate their peak oxygen consumption. Participants will then undergo a maximal cardiopulmonary exercise test (CPET), where peak oxygen consumption will be measured. The Seismofit estimated peak oxygen consumption will be compared with CPET measured peak oxygen consumption (unless prespecified criteria for a maximal exercise test are not met).
  Interventions: Device: Seismofit

INTERVENTIONS:
Device: Seismofit — The Seismofit device uses seismocardiography to estimate peak oxygen consumption from a resting measurement. This study will assess its validity against the gold standard measure of peak oxygen consumption, cardiopulmonary exercise test, conducted as part of standard care.

SUMMARY:
Physical fitness levels of people waiting for a planned operation are often measured using an exercise test. This is because fitness levels help doctors make a plan to improve each person's chances of a successful recovery after their planned operation. The exercise test requires skilled staff, expensive equipment, a 1 hour appointment, and the patient to exercise heavily during the test.

Ventriject, a small to medium sized enterprise, have designed a device called Seismofit that estimates fitness levels of people from a measurement taken whilst laying down. It measures the vibrations of the chest wall caused by the beating heart and uses this information with additional information, such as height, weight and sex, to estimate fitness. The measurement takes around 5 minutes to perform, does not require heavy exercise, expensive equipment or skilled staff.

The Seismofit device was shown to be accurate in young fairly fit people. It has not been tested in people who undergo an exercise test before an operation, who are less fit on average compared to the people that the device was originally tested on. It is likely that the calculations used to estimate fitness levels with the Seismofit device will need to be adjusted for people waiting for an operation. There are two parts to this study. The first part aims to estimate up to 50 people's fitness with the Seismofit device and use directly measured fitness from their standard exercise test before their operation to adjust the calculations for estimating fitness. The second part of this study aims to have a further 50 people undergo the Seismofit device measurement and compare the estimated fitness level with the results from the standard exercise test before an operation. This is to see if the Seismofit device is valid at estimating fitness in people awaiting surgery.

ELIGIBILITY:
Inclusion:

* Adults awaiting major or complex elective surgery classified by the NICE NG45 guideline
* Referred for and capable of performing a maximum effort CPET as part of standard care within their preoperative assessment
* Able to be fully supine for 5 minutes

Exclusion:

* Pacemaker, implantable defibrillator, or any other implantable electronic device in situ
* Permanent Atrial fibrillation, or other persistent arrhythmia (such as, atrial flutter, bigeminy, trigeminy, frequent premature atrial/ventricular complexes, 2nd degree heart block) documented in the patient's medical history
* Body mass index (BMI) >35 kg.m-2
* Severe COPD (defined as FEV1 % predicted <50% [GOLD report, 2022])
* Pectus excavatum or other chest wall deformity
* Claudication that limits exercise tolerance
* Unable to perform maximal CPET
* Refusal to give informed consent
* Presence of an absolute contraindication to CPET detailed in the POETTS clinical guideline (Levett et al. 2018).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1 outcome - refine algorithm | Up to 6 months
  Up to 50 patients awaiting major surgery will have their estimated V̇O2peak (ml/kg/min) recorded using the Seismofit device and actual V̇O2peak (ml/kg/min) measured in their standard preoperative cardiopulmonary exercise test. The Seismofit algorithm will be adjusted using these data points with machine learning.
Phase 2 outcome - validity of refined algorithm | 12 months
  The correlation between the new seismofit algorithm estimate of V̇O2peak (ml/kg/min) and CPET measured and verified V̇O2peak (ml/kg/min) in up to 50 preoperative patients that have valid tests in accordance with maximal exercise test criteria stated in the protocol (RER > 1.10 or maximum heart rate attained within 10 beats of predicted maximum).

SECONDARY OUTCOMES:
Bland-Altman analysis | 12 months
  Agreement between Seismofit estimated V̇O2peak (ml/kg/min) and CPET measured V̇O2peak (ml/kg/min) using Bland-Altman analysis.
Existing V̇O2peak predicted equation analysis | 12 months
  To calculate the correlation and agreement between existing equations used to predict V̇O2peak (ml/kg/min) with directly measured V̇O2peak (ml/kg/min) to observe how these data compare with the Seismofit correlation and agreement data.

OTHER OUTCOMES:
Seismofit total population analysis | 12 months
  Correlation between Seismofit estimated V̇O2peak (ml/kg/min) and CPET measured V̇O2peak (ml/kg/min), including patients that did not meet maximum effort criteria for CPET (RER >1.10 or <10 beats/min estimated maximum heart rate).

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - York and Scarborough NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: No